CLINICAL TRIAL: NCT05096039
Title: Role of Sacubitril/Valsartan in Improving Provider Performance in Managing Heart Failure Under Medicare Alternative Payment Models
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CLCZ696BUS29
Record Dates: First submitted 2021-09-27; First posted 2021-10-27 (Actual); Last update posted 2021-12-16 (Actual); Status verified 2021-12

CONDITIONS: Heart Failure
Keywords: Heart failure,; Medicare,; Alternative Payment Models,; HFrEF,; Healthcare Expenditures
MeSH Terms: conditions — Heart Failure | interventions — sacubitril and valsartan sodium hydrate drug combination; Angiotensin-Converting Enzyme Inhibitors; Valsartan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Treatment Group 1 (use of sacubitril/valsartan): Beneficiaries with one or more prescription claim with an NDC for sacubitril/valsartan during the 90-day episode window (for BPCA) and CY2018 (for MSSP). Patients who met these criteria were assigned a value of '1'; patients that did not meet these criteria were assigned a value of '0'
  Interventions: Drug: Sacubitril/valsartan
- Treatment Group 2 (use of ACEI or ARB and no use of sacubitril/valsartan): Beneficiaries with one or more prescription claim with an NDC for any ACEI/ARB and no prescription claims for sacubitril/valsartan during the 90-day episode window (for BPCA) and CY2018 (for MSSP). Patients who met these criteria were assigned a value of '1'; patients that did not meet these criteria were assigned a value of '0'
  Interventions: Drug: ACEI or ARB and no sacubitril/valsartan
- Treatment Group 3 (no use of ACEI, ARB, or sacubitril/valsartan): Beneficiaries who did not qualify for Group 1 or Group 2 were assigned a value of '1'; patients that did not meet this criteria were assigned a value of '0'
- Cohort Group 1 (Overall cohort): The beneficiaries who met the inclusion criteria and were divided into the three treatment groups were considered Cohort Group 1 or the "overall cohort."
- Cohort Group 2 (subgroup 1): Patients with evidence of systolic HF defined as: having at least 2 medical claims (on different dates) with an ICD-9/-10 diagnosis code for systolic HF in any position during the lookback period and/or during the entire 90-day episode window (for BPCA) and CY2017 and/or CY2018 (for MSSP). Patients who met these criteria were assigned a value of '1'; patients that did not meet these criteria were assigned a value of '0'
- Cohort Group 3 (subgroup 2): Patients with evidence of Heart Failure Reduced Ejection Fraction (HFrEF) identified based on a published algorithm

INTERVENTIONS:
Drug: Sacubitril/valsartan — Beneficiaries with one or more prescription claim with an NDC for sacubitril/valsartan (from the PDE file) during the 90-day episode window. Patients who met these criteria were assigned a value of '1'; patients that did not meet these criteria were assigned a value of '0'
  Groups: Treatment Group 1 (use of sacubitril/valsartan)
Drug: ACEI or ARB and no sacubitril/valsartan — Beneficiaries with one or more prescription claim with an NDC for any ACEI/ARB and no prescription claims for sacubitril/valsartan during the 90-day episode window. Patients who met these criteria were assigned a value of '1'; patients that did not meet these criteria were assigned a value of '0'
  Groups: Treatment Group 2 (use of ACEI or ARB and no use of sacubitril/valsartan)

SUMMARY:
This study evaluated the association between sacubitril/valsartan utilization and HF patients' Part A & B expenditures within the reimbursement framework of BPCI and MSSP, and identified BPCI/MSSP participants with the greatest potential for performance improvement (with respect to improving quality and efficiency of care for HF patients) through optimized utilization of sacubitril/valsartan.

DETAILED DESCRIPTION:
This drug utilization study employed a retrospective cohort design using the 100% files of 2015-2018 Medicare enrollment and Part A, B & D claims data in conjunction with publicly available information on providers participating in Bundled Payments for Care Improvement (BPCI) and/or Medicare Shared Savings Program (MSSP).

BPCI Study Design The unit of analysis for addressing study objectives was a unique Congestive Heart Failure (CHF) episode of care, which encompassed an initial acute inpatient stay plus all Part A & B covered medical services during the 90 days post hospital discharge. Episode index date was defined as the date of a beneficiary's initial acute hospital stay with a qualifying Medicare Severity-Diagnosis Related Group (MS-DRG) for CHF, triggering a CHF episode of care. Beneficiaries were followed longitudinally from episode index date through episode end date to measure their utilization of sacubitril/valsartan and Part A & B expenditures during the CHF episode of care. A 12-month lookback period, based on when the episode was initiated, was utilized to capture beneficiaries' baseline characteristics. For example, episodes initiated on 2/1/2018 will have a 2/1/2017 to 1/31/2018 baseline lookback period. Balancing the need for data recency, all qualifying CHF episodes from 2016-2018 were included in the analysis. Given this is an episode-level analysis, a beneficiary may have contributed multiple CHF episodes to the data analysis. To account for potential within-subject clustering, a generalized linear model with a gamma distribution was applied for estimating the association between sacubitril/valsartan use and CHF episode costs.

MSSP Study Design The unit of analysis for addressing study objectives was a HF patient's Part A & B expenditures within the MSSP. Given the most recent year of data available at the time the study was conducted was 2018, the study population included HF patients for whom the MSSP participants were accountable in 2018 per Centers for Medicare & Medicaid Services (CMS) assignment. These beneficiaries' utilization of sacubitril/valsartan and annual Part A & B expenditures was measured from January 1, 2018 - December 31, 2018. Data from CY 2017 was leveraged for capturing these patients' baseline characteristics.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old during year of index date with valid gender and geographic information
* Continuous enrollment (CE) in the health plan with medical and pharmacy benefits for ≥6 months (180ii days) before the index date (pre-index period)
* CE with medical and pharmacy benefits for ≥18 months (540ii days) beginning on the index date (post-index period)
* All patients had uniform 6-month pre-index and 18-month post-index periods
* ≥1 medical claim with an MS diagnosis codeiii in any position during the pre-or post-index periods
* ≥1 claim for fingolimod after the index date (i.e., from index date +1 to 539 days post-index)
* By requiring ≥1 medical claim with an MS diagnosis code and ≥2 claims with an NDC for fingolimod, the inclusion criteria essentially incorporated the preferred/overall best performing MS case-finding definition validated by Culpepper et al. The criteria for that definition required at least 3 separate encounters from any of the following: MS-related ambulatory visits, MS-related inpatient stays, and DMT claims during a 12-month period. Slightly higher accuracy was found when a 24-month period was used.

Exclusion criteria

≥1 pharmacy or medical claim for any MS DMT during the pre-index period

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult Medicare FFS beneficiaries diagnosed with HF and who received care from a BPCI or MSSP participant
Sampling Method: Probability Sample
Enrollment: 1614719 (Actual)
Dates: Start 2020-04-10 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Bundled Payments for Care Improvement (BPCI) Congestive Heart Failure (CHF) episode costs | 90 days following the episode index date (episode index date differed by patient depending on when they were admitted to the hospital (triggering a HF clinical episode), ranging from Jan. 1, 2016 through Oct. 1, 2018)
  BPCI CHF episode costs defined as the sum of expenditures for Part A & B covered medical services during the CHF episode

SECONDARY OUTCOMES:
Medicare Shared Savings Program (MSSP) beneficiary annual Medicare | Baseline (Calender Year 2017) and Calender Year 2018 (01/01/2018 to 31/12/2018)
  MSSP beneficiary annual Medicare Part A & B expenditures defined as the sum of all Part A & B expenditures within the calendar year (CY)
Outpatient utilization of sacubitril/valsartan during 90-day post-discharge period of the CHF episode | 90 days following the episode index date (episode index date differed by patient depending on when they were admitted to the hospital (triggering a HF clinical episode), ranging from Jan. 1, 2016 through Oct. 1, 2018)
  yes/no binary variable
Difference in actual Congestive Heart Failure (CHF) episode costs vs. benchmark CHF episode costs | 90 days following the episode index date (episode index date differed by patient depending on when they were admitted to the hospital (triggering a HF clinical episode), ranging from Jan. 1, 2016 through Oct. 1, 2018)
  A benchmark was created to assess performance and determine savings for the BPCI. Difference in actual Congestive Heart Failure (CHF) episode costs vs. benchmark CHF episode costs were reported
Outpatient utilization of sacubitril/valsartan among Medicare Shared Savings Program (MSSP) Heart Failure (HF) patients | Baseline (Calender Year 2017) and Calender Year 2018 (01/01/2018 to 31/12/2018)
  yes/no binary variable
Difference in actual HF patient annual Medicare Part A & B expenditures vs. benchmark HF patient annual Medicare Part A & B expenditures | Baseline (Calender Year 2017) and Calender Year 2018 (01/01/2018 to 31/12/2018)
  A benchmark was created to assess performance and determine savings for the MSSP. Difference in actual HF patient annual Medicare Part A & B expenditures vs. benchmark HF patient annual Medicare Part A & B expenditures were reported

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Pharmaceuticals, East Hanover, New Jersey, United States

REFERENCES:
- See also: Results for CLCZ696BUS29 from the Novartis Clinical Trials Website — http://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17867